CLINICAL TRIAL: NCT03968575
Title: The Affiliated Eye Hospital of Wenzhou Medical University
Brief Title: Sub-threshold Micro-Pulse Laser Therapy for Drusen of Dry AMD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Eye Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Xiaoling Liu, Clinical Professor, The Eye Hospital of Wenzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-075-K-74
Record Dates: First submitted 2019-05-22; First posted 2019-05-30 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Drusen
MeSH Terms: interventions — Laser Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laser (Experimental)
  Interventions: Device: laser treatment

INTERVENTIONS:
Device: laser treatment — sub-threshold micro-pulse laser treatment

SUMMARY:
To investigate the efficacy and safety of sub-threshold micro-pulse laser therapy for drusen of dry age-related macular degeneration (AMD) .

ELIGIBILITY:
Inclusion Criteria:

1. Older than 50 years of age.
2. Male or female patients with nonexudative AMD with a drusen diameter of at least 125um in the central 3mm circle
3. clear media to perform colour, red-free imaging and fundus fluorescein angiography, fundus autofluorescence imaging and OCT.
4. Able to give an informed consent.

Exclusion Criteria:

1. Presence of other macular disease such as epiretinal membrane, macular telangiectasia.
2. unclear media that no clear colour, red-free imaging and fundus fluorescein angiography, fundus autofluorescence imaging and OCT can performed.
3. Ocular or periocular infections.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in macular drusen volume | 6 and 12 months
  Mean change in macular drusen volume on optical coherence tomograph(OCT)
Change in macular drusen area | 6 and 12 months
  Mean change in macular drusen area on OCT

SECONDARY OUTCOMES:
Change in visual acuity | 6 and 12 months
  Mean change in best-corrected visual acuity

CONTACTS AND LOCATIONS:
Locations (1):
- The eye of Wenzhou Medical University, Wenzhou, Zhejiang, China